CLINICAL TRIAL: NCT01582789
Title: Clinical Evaluation of CooperVision's Avaira Spherical Daily Wear Soft Contact Lens Versus Vistakon's Oasys Spherical Daily Wear Soft Contact Lens
Brief Title: Comparative Study of Two Marketed Spherical Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-37
Record Dates: First submitted 2012-04-12; First posted 2012-04-23 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- enfilcon A/senofilcon A (Active Comparator): Subjects were randomized to wear enfilcon A then Senofilcon A for two weeks.
  Interventions: Device: enfilcon A; Device: senofilcon A
- senofilcon A/enfilcon A (Active Comparator): Subjects were randomized to wear senofilcon A then enfilcon A for two weeks
  Interventions: Device: enfilcon A; Device: senofilcon A

INTERVENTIONS:
Device: enfilcon A — enfilcon A daily wear soft contact lens
Device: senofilcon A — senofilcon A daily wear soft contact lens

SUMMARY:
The purpose of this study is to obtain objective and subjective clinical data to compare the performance of two soft contact lenses.

DETAILED DESCRIPTION:
The study will evaluate the daily wear performance of the Avaira (enfilcon A) spherical lens during two weeks of wear compared to Vistakon's Oasys (senofilcon A) spherical lens.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following conditions prior to inclusion in the study:

* Based on his/her knowledge, must be in good general health.
* Be 18 to 38 years old.
* Be able and willing to adhere to the instructions set forth in this protocol and complete all specified evaluation.
* Read, indicate understanding of, and sign Written Informed Consent.
* Be existing or successfully adapted users of soft contact lenses, but not currently wearing either of the study lenses being evaluated in this trial.
* Require a visual correction in both eyes.
* Require a prescription between +8.00D and -12.00D and have less than -0.75D of astigmatism in both eyes.
* Achieve visual acuity of 20/25 or better in each eye with a spherical contact lens prescription.
* Must be able to wear their lenses at least 10 working days over the next 2-weeks; > 8 hours/day assuming there are no contraindications for doing so.
* Have normal eyes with no evidence of abnormality or disease. For the purposes of this study a normal eye is defined as one having: no amblyopia; no evidence of lid abnormality or infection (e.g. entropion, ectropion, chalazia, recurrent styes); no clinically significant slit lamp findings (e.g. infiltrates or other slit lamp findings Grade 2 or above: corneal edema, tarsal abnormalities, and conjunctival injection); no other active ocular disease (e.g. glaucoma, history of recurrent corneal erosions, cornea [infiltrates], conjunctiva, lids, and intraocular infection or inflammation of an allergic, bacterial, or viral etiology); no aphakia

Exclusion Criteria:

Any of the following will render a subject ineligible for inclusion:

* Greater than 0.50D of refractive astigmatism in either eye.
* Presbyopic or current monovision contact lens wear.
* Cannot be currently wearing of either lenses (Avaira or Oasys)
* Presence of clinically significant (grade 2-4) anterior segment abnormalities; inflammations such as iritis; or any infection of the eye, lids, or associated structures.
* Presence of ocular or systemic disease or need of medication which might interfere with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear such as: pathological dry eye or associated findings; pterygium, pinguecula or corneal scars within the visual axis; neovascularization > 0.75 mm in from the limbus, giant papillary conjunctivitis (GPC) worse than Grade 1; anterior uveitis or iritis (past or present), seborrheic eczema, seborrheic conjunctivitis, history of corneal ulcer or fungal infections; poor personal hygiene
* A known history of corneal hypoesthesia (reduced corneal sensitivity).
* Contact lens best corrected Snellen visual acuities (VA) worse than 20/30.
* Aphakia, Keratoconus or a highly irregular cornea

To be eligible to enter the study, subjects must have ALL of the inclusion criteria and NONE of the exclusion criteria present.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2012-04-09; Primary Completion 2012-05 (Actual); Study Completion 2012-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Siegel, OD, Study Director — CooperVision, Inc.
Locations (2):
- United States (2):
  - Advanced Eyecare, Pismo Beach, California
  - Eric M. White, OD, Inc., San Diego, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Enfilcon A, Then Senofilcon A: Subjects were randomized to wear enfilcon A then Senofilcon A for two weeks
  enfilcon A: enfilcon A daily wear soft contact lens
  senofilcon A: senofilcon A daily wear soft contact lens
- Senofilcon A, Then Enfilcon A: Subjects were randomized to wear senofilcon A then enfilcon A for two weeks
  senofilcon A: senofilcon A daily wear soft contact lens
  enfilcon A: enfilcon A daily wear soft contact lens
Period: First Intervention (14 Days)
Arm/Group | Enfilcon A, Then Senofilcon A | Senofilcon A, Then Enfilcon A
Started | 34 | 27
Completed | 34 | 27
Not Completed | 0 | 0
Period: Second Intervention (14 Days)
Arm/Group | Enfilcon A, Then Senofilcon A | Senofilcon A, Then Enfilcon A
Started | 34 | 27
Completed | 33 | 27
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects prior to dispense of first set of study lenses
Groups:
- Overall Study Group Prior to Dispense: All subjects prior to dispense of first set of study lenses
Arm/Group | Overall Study Group Prior to Dispense
Number analyzed (Participants) | 61
Age, Continuous [Median (Full Range); unit: years] | 30 [19 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Comfort - First Intervention
Description: Comfort - on insertion and overall assessed at baseline for first intervention on a scale 0-10. 0=uncomfortable/cannot tolerate, 10=very comfortable/cannot be felt,
Time Frame: Baseline
Population: one drop out at first 2 week follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enfilcon A: Subject wears enfilcon A daily wear soft contact lens as first pair
- Senofilcon A: Subject wears senofilcon A daily wear soft contact lens as first pair
Arm/Group | Enfilcon A | Senofilcon A
Number analyzed (Participants) | 34 | 27
units on a scale
  Insertion | 9.3 (1.1) | 9.3 (1.1)
  Overall | 9.4 (0.9) | 9.3 (0.9)

2. Primary Outcome: Comfort - Second Intervention
Description: as for outcome 1
Time Frame: Baseline
Population: one drop out at first 2 week follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enfilcon A: Subject wears enfilcon A daily wear soft contact lens as second pair
- Senofilcon A: Subject wears senofilcon A daily wear soft contact lens as second pair
Arm/Group | Enfilcon A | Senofilcon A
Number analyzed (Participants) | 27 | 33
units on a scale
  Insertion | 9.1 (1.1) | 9.1 (1.3)
  Overall | 9.1 (1.0) | 9.1 (0.9)

3. Primary Outcome: Comfort - First Intervention
Description: Participant response of comfort for first intervention of study lenses assessed at 2 weeks. Comfort at insertion, comfort at end of day, comfort at 2 weeks, and overall comfort were rated on subjective response scale. (Scale 0-10, 0=uncomfortable/cannot tolerate, 10=very comfortable/cannot be felt).
Time Frame: 2 Weeks
Population: one drop out at first 2 week follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enfilcon A | Senofilcon A
Number analyzed (Participants) | 34 | 27
units on a scale
  Insertion | 8.5 (1.8) | 8.3 (2.0)
  End of day | 7.2 (2.1) | 7.7 (1.7)
  2 weeks wear | 7.7 (2.0) | 7.7 (2.1)
  Overall | 7.9 (1.7) | 8.2 (1.8)

4. Primary Outcome: Comfort - Second Intervention
Description: as for outcome 3
Time Frame: 2 Weeks
Population: 1 subject withdrew from study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enfilcon A | Senofilcon A
Number analyzed (Participants) | 27 | 33
units on a scale
  Insertion | 8.5 (1.1) | 8.4 (1.6)
  End of day | 6.3 (2.2) | 7.1 (2.3)
  2 weeks wear | 7.4 (1.8) | 7.3 (2.4)
  Overall | 7.2 (1.8) | 7.6 (2.4)

5. Primary Outcome: Comfortable Wearing Time - First Intervention
Description: Comfortable Wearing Time. (Participant response in number of hours) Obtained at 2 weeks wear for first intervention at week two visit.
Time Frame: 2 Weeks
Population: one drop out at first 2 week follow up
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Enfilcon A | Senofilcon A
Number analyzed (Participants) | 33 | 27
hours | 11.5 (3.5) | 10.7 (3.2)

6. Primary Outcome: Comfortable Wearing Time - Second Intervention
Description: Comfortable Wearing Time. (Participant response in number of hours) Obtained at 2 weeks wear for second intervention at week two visit.
Time Frame: 2 Weeks
Population: one drop out at first 2 week follow up
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Enfilcon A | Senofilcon A
Number analyzed (Participants) | 27 | 33
hours | 10.1 (3.0) | 11 (3.9)

ADVERSE EVENTS:
Time Frame: From dispense up to 2 weeks for each intervention
Groups:
- Enfilcon A/Senofilcon A: enfilcon A daily wear soft contact lens 1st then cross over and subject wears the senofilcon A daily wear soft contact lens 2nd
  enfilcon A: enfilcon A daily wear soft contact lens
  senofilcon A: senofilcon A daily wear soft contact lens
- Senofilcon A/Enfilcon A: senofilcon A daily wear soft contact lens 1st then cross over and subject wears the enfilcon A daily wear soft contact lens 2nd
  enfilcon A: enfilcon A daily wear soft contact lens
  senofilcon A: senofilcon A daily wear soft contact lens
Arm/Group | Enfilcon A/Senofilcon A | Senofilcon A/Enfilcon A
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/27
Other Adverse Events (participants affected / at risk) | 0/34 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor. Assuming that the product is marketed, it is the intention of the sponsor to publish the results of the study.